CLINICAL TRIAL: NCT03862131
Title: PROactive Evaluation of Function to Avoid CardioToxicity
Acronym: PROACT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient funding/staff
Sponsor: Washington University School of Medicine (Other)
Collaborators: Myocardial Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201809177
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cardiotoxicity; Breast Cancer; Lymphoma; Sarcoma; Leukemia; Myeloma; Lung Cancer
MeSH Terms: conditions — Cardiotoxicity; Breast Neoplasms; Lymphoma; Sarcoma; Leukemia; Neoplasms, Plasma Cell; Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Patients will be classified based on baseline segmental MyoStrain Fast-SENC strain testing, into lower and higher risk groups. The higher risk group will be randomized with half blinded and half unblinded to intramyocardial strain in terms of assessing cardiotoxicity incidence and management. Physicians will have knowledge of MyoStrain intramyocardial strain and cardiac MRI information in the unblinded group to augment standard of care in detecting and managing cardiotoxicity. Physicians will not have access to or knowledge of intramyocardial strain and cardiac MRI data, except 4 standard cardiac measures, for patients in the blinded group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MyoStrain® unblinded treatment arm (Experimental): * After consenting to the PROACT study, patients will undergo a baseline MRI to determine their risk stratification for the study. This baseline MyoStrain® MRI must demonstrate 2 or more segments measuring >-10% or 9 or more segments >-17% for entrance into the study as the Higher Risk Group
  * The unblinded treatment arm will enhance patient management by augmenting standard of care with serial MyoStrain® monitoring of the impact of cancer therapy on myocardial function.
  * Higher Risk unblinded patients will continue to undergo MyoStrain® MRI testing, regardless of study arm, at 1 month (+1 week), 3 months (+ 1 week), 6 months (+1 week), 12 months (+ 30 days), 24 months (+30 days), and 36 months (+30 days) after the baseline visit.
  * In addition to the MyoStrain® testing, patients will also be asked to complete a brief patient satisfaction questionnaire at each PROACT time point.
  Interventions: Device: MyoStrain®
- MyoStrain® blinded control arm (Active Comparator): * After consenting to the PROACT study, patients will undergo a baseline MRI to determine their risk stratification for the study. This baseline MyoStrain® MRI must demonstrate 2 or more segments measuring >-10% or 9 or more segments >-17% for entrance into the study as the Higher Risk group
  * The blinded control arm will provide investigators with LVEF and LVEDV/LVESV measurements, which are clinical, in conjunction with standard of care
  * Higher Risk blinded patients will continue to undergo MyoStrain® MRI testing, regardless of study arm, at 1 month (+1 week), 3 months (+ 1 week), 6 months (+1 week), 12 months (+ 30 days), 24 months (+30 days), and 36 months (+30 days) after the baseline visit.
  * In addition to the MyoStrain® testing, patients will also be asked to complete a brief patient satisfaction questionnaire at each PROACT time point.
  Interventions: Device: MyoStrain®

INTERVENTIONS:
Device: MyoStrain® — MyoStrain® SENC software receives image data from MRI storage archives and performs viewing, image manipulation, communication, printing, and quantification of images.
  Other Names: Cardiac MRI Imaging Software; Intramyocardial Strain

SUMMARY:
This study is intended to evaluate the ability of an intramyocardial strain analysis package with cardiac MRI to assist in the early detection and management of cardiotoxicity from therapeutics used to treat cancer.

DETAILED DESCRIPTION:
The primary purpose of the PROACT study is to test the accuracy of MyoStrain® to detect cardiotoxicity in patients on high risk cancer therapy. After undergoing baseline MRI and meeting eligibility criteria, patients will be further randomized to an unblinded arm (MyoStrain® measured and available to the treatment team) and a blinded arm (MyoStrain® measured but not available to the treatment team). This randomization will aid in an exploratory aim of testing the feasibility of MyoStrain® to guide cardioprotective therapy in the unblinded vs blinded arms. However, as all patients will have MyoStrain® measured, all patients (both treatment arms) will be combined for testing the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the SURVIVE registry
* Signed informed consent form for PROACT
* Histological diagnosis of any cancer type (patients with treated and clinically stable brain metastasis are acceptable)
* Scheduled to receive anti-cancer therapy (radiation therapy is permitted)

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI)
* Unable to comply with study investigations (in the judgment of the investigator)
* Life expectancy less than 1 year
* Note: If a patient develops a temporary contraindication (e.g. temporary tissue expanders in breast cancer patients) after the baseline MRI, follow up MRIs will be discontinued for safety for the duration in which the patient has the contraindication. However, once the patient is no longer contraindicated to receiving MRIs, the study schedule may resume with their next scheduled MRI time point from the date of enrollment. Therefore, some time points may be skipped during the patient's enrollment in the study.

Also, if a patient needs a repeat MRI at any time point for any reason (i.e. panic attack during the MRI causing them to not be able to continue, unreadable images, etc.), we may repeat the MRI as long as the patient is willing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Mitchell, M.D., MSCI, FACC, FICOS, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Daniel J. Lenihan, Gregory M. Lanza, Pamela K. Woodard, Joshua Mitchell, SUPERIOR DETECTION OF CARDIOTOXICITY USING CARDIAC MRI MYOSTRAIN DURING CANCER CHEMOTHERAPY, Journal of the American College of Cardiology, Volume 83, Issue 13, Supplement, 2024, Page 2350, ISSN 0735-1097, https://doi.org/10.1016/S0735-1097(24)04340-7. (https://www.sciencedirect.com/science/article/pii/S0735109724043407)
- [Result] Joshua Mitchell, Syed Z. Qamer, Gregory M. Lanza, Pamela K. Woodard, JAMES WHAYNE, Daniel J. Lenihan, MYOCARDIAL STRAIN GUIDED CARDIOPROTECTION DURING CHEMOTHERAPY WITH CARDIAC MRI IMPROVES CARDIAC HEALTH, Journal of the American College of Cardiology, Volume 83, Issue 13, Supplement, 2024, Page 2673, ISSN 0735-1097, https://doi.org/10.1016/S0735-1097(24)04663-1. (https://www.sciencedirect.com/science/article/pii/S0735109724046631)
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-randomized: -Patients were enrolled but not randomized to either arm.
Period: Overall Study
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Non-randomized
Started | 25 | 18 | 6
Completed | 15 | 10 | 0
Not Completed | 10 | 8 | 6
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Determined to be ineligible | 0 | 0 | 5
Not completed — Death | 4 | 4 | 0
Not completed — Withdrawal by Subject | 5 | 3 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Non-randomized | Total
Number analyzed (Participants) | 25 | 18 | 6 | 49
Age, Continuous [Median (Full Range); unit: years] | 55 [26 to 72] | 58.5 [21 to 73] | 48.5 [39 to 67] | 55 [21 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 11 | 5 | 36
  Male | 5 | 7 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 17 | 6 | 48
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 1 | 5
  White | 21 | 18 | 5 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 18 | 6 | 49

OUTCOME MEASURES:

1. Primary Outcome: ROC AUC of MyoStrain® Compared to Standard CMR Measurements (LV End Diastolic Volume Index, LV End Systolic Volume Index, LV Stroke Volume Index and Left Ventricular Ejection Fraction) to Detect Myocardial Dysfunction During Cancer Treatment
Description: The area under the curve refers to the area under the curve of Receiver operating characteristic curves (ROC AUC) to evaluate the accuracy of MyoStrain® to detect cardiotoxicity compared to Cardiovascular Magnetic Resonance (CMR) Imaging standard measurements.
  * Myocardial dysfunction was defined as the occurrence of either clinical or subclinical cardiotoxicity.
  * Clinical cardiotoxicity was defined as an absolute change in LVEF > 10% from baseline to below 53% combined with heart failure symptoms or elevation in NT pro BNP to above 199 pg/mL.
  * In patients with LVEF < 53% at baseline, clinical cardiotoxicity was defined by a symptomatic drop in LVEF > 10% or a HF hospitalization.
  * Subclinical CTX was defined as an asymptomatic patient with a greater than 10% decrease in LVEF, worsening GLS more than 15% from baseline, or new elevation in NT pro BNP >199 pg/mL.
Time Frame: Through 36 months
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Combined MyoStrain® Control Arm and Treatment Arm: * After consenting to the PROACT study, patients will undergo a baseline MRI to determine their risk stratification for the study. This baseline MyoStrain® MRI must demonstrate 2 or more segments measuring >-10% or 9 or more segments >-17% for entrance into the study as the Higher Risk Group.
  * After meeting eligibility criteria, patients will be further randomized to an unblinded arm (MyoStrain® measured and available to the treatment team) and a blinded arm (MyoStrain® measured but not available to the treatment team). This randomization will aid in an exploratory aim of testing the feasibility of MyoStrain® to guide cardioprotective therapy in the unblinded vs blinded arms. However, as all patients will have MyoStrain® measured, all patients (both treatment arms) will be combined for testing the primary outcome measure.
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Combined MyoStrain® Control Arm and Treatment Arm
Number analyzed (Participants) | 25 | 18 | 43
probability
  MyoStrain® | 0.876 [0.770 to 0.982] | 0.853 [0.728 to 0.978] | 0.864 [0.783 to 0.946]
  CMR LVEF | 0.603 [0.456 to 0.749] | 0.790 [0.648 to 0.933] | 0.679 [0.573 to 0.786]
  CMR left ventricular end-diastolic indexed (LVEDVI) | 0.522 [0.377 to 0.666] | 0.532 [0.370 to 0.693] | 0.515 [0.408 to 0.622]
  CMR left ventricular end-systolic volume index (LVESVI) | 0.501 [0.358 to 0.645] | 0.689 [0.531 to 0.847] | 0.589 [0.481 to 0.698]
  CMR left ventricular stroke volume index (LVSVI) | 0.574 [0.428 to 0.721] | 0.693 [0.535 to 0.850] | 0.627 [0.519 to 0.735]

2. Primary Outcome: Sensitivity of MyoStrain® Compared to CMR Standard Measurements (LV End Diastolic Volume Index, LV End Systolic Volume Index, LV Stroke Volume Index and Left Ventricular Ejection Fraction) to Detect Myocardial Dysfunction During Cancer Treatment
Description: Sensitivity is defined as the number of true positives divided by the number of true positives + number of false negatives.
  * Myocardial dysfunction was defined as the occurrence of either clinical or subclinical cardiotoxicity.
  * Clinical cardiotoxicity was defined as an absolute change in LVEF > 10% from baseline to below 53% combined with heart failure symptoms or elevation in NT pro BNP to above 199 pg/mL.
  * In patients with LVEF < 53% at baseline, clinical cardiotoxicity was defined by a symptomatic drop in LVEF > 10% or a HF hospitalization.
  * Subclinical CTX was defined as an asymptomatic patient with a greater than 10% decrease in LVEF, worsening GLS more than 15% from baseline, or new elevation in NT pro BNP >199 pg/mL
Time Frame: Through 36 months
Measure: Number (95% Confidence Interval); unit: percent sensitivity
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Combined MyoStrain® Control Arm and Treatment Arm
Number analyzed (Participants) | 25 | 18 | 43
percent sensitivity
  MyoStrain® | 83.3 [66.1 to 100.0] | 66.7 [42.8 to 90.5] | 84.8 [78.3 to 94.6]
  CMR LVEF | 33.3 [11.6 to 55.1] | 53.3 [28.1 to 78.6] | 42.4 [25.6 to 59.3]
  CMR left ventricular end-diastolic indexed (LVEDVI) | 44.4 [21.5 to 67.4] | 66.7 [42.8 to 90.5] | 48.5 [31.4 to 65.5]
  CMR left ventricular end-systolic volume index (LVESVI) | 22.2 [3.0 to 41.4] | 66.7 [42.8 to 90.5] | 45.5 [28.5 to 62.4]
  CMR left ventricular stroke volume index (LVSVI) | 33.3 [11.6 to 55.1] | 93.3 [80.7 to 100.0] | 33.3 [17.2 to 49.4]

3. Primary Outcome: Specificity of MyoStrain® and CMR Standard Measurements (LV End Diastolic Volume Index, LV End Systolic Volume Index, LV Stroke Volume Index and Left Ventricular Ejection Fraction) to Detect Myocardial Dysfunction During Cancer Treatment
Description: Specificity is defined as the number of true negatives divided by the number of true negatives + number of false positives.
  * Myocardial dysfunction was defined as the occurrence of either clinical or subclinical cardiotoxicity.
  * Clinical cardiotoxicity was defined as an absolute change in LVEF > 10% from baseline to below 53% combined with heart failure symptoms or elevation in NT pro BNP to above 199 pg/mL.
  * In patients with LVEF < 53% at baseline, clinical cardiotoxicity was defined by a symptomatic drop in LVEF > 10% or a HF hospitalization.
  * Subclinical CTX was defined as an asymptomatic patient with a greater than 10% decrease in LVEF, worsening GLS more than 15% from baseline, or new elevation in NT pro BNP > 199 pg/mL
Time Frame: Through 36 months
Measure: Number (95% Confidence Interval); unit: percent specificity
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Combined MyoStrain® Control Arm and Treatment Arm
Number analyzed (Participants) | 25 | 18 | 43
percent specificity
  MyoStrain® | 77.9 [70.5 to 85.2] | 88.4 [81.6 to 95.1] | 73.6 [67.6 to 79.6]
  CMR LVEF | 95.0 [91.2 to 98.9] | 90.5 [84.2 to 96.8] | 86.3 [81.6 to 91.0]
  CMR left ventricular end-diastolic indexed (LVEDVI) | 75.2 [67.5 to 82.9] | 52.4 [41.7 to 63.1] | 61.5 [54.8 to 68.1]
  CMR left ventricular end-systolic volume index (LVESVI) | 99.2 [97.6 to 100.0] | 69.0 [59.2 to 78.9] | 76.6 [70.8 to 82.4]
  CMR left ventricular stroke volume index (LVSVI) | 92.6 [87.9 to 97.2] | 42.9 [32.3 to 55.4] | 90.7 [86.8 to 94.7]

4. Primary Outcome: Accuracy of MyoStrain® and CMR Standard Measurements (LV End Diastolic Volume Index, LV End Systolic Volume Index, LV Stroke Volume Index and Left Ventricular Ejection Fraction) to Detect Myocardial Dysfunction During Cancer Treatment
Description: Accuracy is defined as (true positives + true negatives) divided by the total number of cases
  * Myocardial dysfunction was defined as the occurrence of either clinical or subclinical cardiotoxicity.
  * Clinical cardiotoxicity was defined as an absolute change in LVEF > 10% from baseline to below 53% combined with heart failure symptoms or elevation in NT pro BNP to above 199 pg/mL.
  * In patients with LVEF < 53% at baseline, clinical cardiotoxicity was defined by a symptomatic drop in LVEF > 10% or a HF hospitalization.
  * Subclinical CTX was defined as an asymptomatic patient with a greater than 10% decrease in LVEF, worsening GLS more than 15% from baseline, or new elevation in NT pro BNP >199 pg/mL.
Time Frame: Through 36 months
Measure: Number (95% Confidence Interval); unit: percent accuracy
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Combined MyoStrain® Control Arm and Treatment Arm
Number analyzed (Participants) | 25 | 18 | 43
percent accuracy
  MyoStrain® | 78.6 [71.8 to 85.4] | 85.1 [78.2 to 92.1] | 75.1 [69.6 to 80.6]
  CMR LVEF | 87.1 [81.5 to 92.6] | 84.8 [77.8 to 91.9] | 80.3 [75.2 to 85.3]
  CMR left ventricular end-diastolic indexed (LVEDVI) | 71.2 [63.7 to 78.7] | 54.5 [44.7 to 64.4] | 59.7 [53.4 to 65.9]
  CMR left ventricular end-systolic volume index (LVESVI) | 89.2 [84.1 to 94.4] | 68.7 [59.6 to 77.8] | 72.3 [66.6 to 78.0]
  CMR left ventricular stroke volume index (LVSVI) | 84.9 [78.9 to 90.8] | 50.5 [40.7 to 60.4] | 82.8 [78.0 to 87.6]

5. Primary Outcome: Independent Effectiveness of MyoStrain® to Detect Cardiac Dysfunction Compared to Standard Cardiac Imaging Measures
Description: Myocardial dysfunction is the occurrence of either clinical or subclinical cardiotoxicity.
  * Clinical cardiotoxicity was defined as an absolute change in LVEF >10% from baseline to below 53% combined with heart failure symptoms or elevation in NT pro BNP to above 199 pg/mL
  * In patients with LVEF <53% at baseline, clinical cardiotoxicity was defined by a symptomatic drop in LVEF >10% or a HF hospitalization
  * Subclinical CTX was defined as an asymptomatic patient with a greater than 10% decrease in LVEF, worsening GLS more than 15% from baseline, or new elevation in NT pro BNP >199 pg/mL
Time Frame: Through 36 months
Population: Events were excluded if there was an earlier event in the same patient closer in time to the MRI scan (6 events). Events were also excluded if they were > 6 months from the last MRI scan (1 event).
Measure: Number; unit: myocardial dysfunction events
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Combined MyoStrain® Control Arm and Treatment Arm
Number analyzed (Participants) | 8 | 10 | 18
myocardial dysfunction events
  Clinical events: number analyzed (Participants) | 4 | 6 | 10
  Clinical events | 7 | 7 | 14
  Subclinical events: number analyzed (Participants) | 7 | 6 | 13
  Subclinical events | 10 | 8 | 18

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality will be tracked from time of consent to the last study visit (up to 36 months).
Description: Only adverse events in relation to the study procedures will be documented and reported. These include adverse events occurring from the MRI scanner, SENC MyoStrain® Testing Software, or breach of confidentiality.
Arm/Group | MyoStrain® Unblinded Treatment Arm | MyoStrain® Blinded Control Arm | Non-randomized
All-Cause Mortality (participants affected / at risk) | 4/25 | 4/18 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 1/25 | 1/18 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MyoStrain® Unblinded Treatment Arm (N=25) | MyoStrain® Blinded Control Arm (N=18) | Non-randomized (N=6)
Anxiety (Psychiatric disorders) | 1 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT03862131/Prot_SAP_000.pdf